CLINICAL TRIAL: NCT04830449
Title: A Multi-center, Randomized, Double-blinded, Active-Controlled, Parallel, Phase III Study to Evaluate the Efficacy and Safety of HCP1904-2 in Essential Hypertension Patients.
Brief Title: Clinical Efficacy and Safety Evaluation of HCP1904-2 in Essential Hypertension Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-CHORUS-302
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Hypertension
Keywords: Losartan; Chlorthalidone
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCP1904-2 (Experimental)
  Interventions: Drug: HCP1904-2
- RLD2001-2 (Active Comparator)
  Interventions: Drug: RLD2001-2

INTERVENTIONS:
Drug: HCP1904-2 — Take it once daily for 8 weeks orally.
  Arms: HCP1904-2
Drug: RLD2001-2 — Take it once daily for 8 weeks orally.
  Arms: RLD2001-2

SUMMARY:
The purpose of this study is to evaluate of efficacy and safety of HCP1904-2 and RLD2001-2 alone in patients with essential hypertension inadequately controlled on RLD2001-2 monotherapy.

DETAILED DESCRIPTION:
A Multi-center, Randomized, Double-blinded, Active-controlled, Parallel, Phse III Study to Evaluate the Efficacy and Safety of HCP1904-2 in Essential Hypertension Patients

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age
2. Patients who understands the process of clinical study and voluntarily signs a peer letter
3. Visit1: A person whose blood pressure measured in visit1 corresponds to the following conditions

   * Blood pressure medication taken patients: 130mmHg ≤ sitSBP<180mmHg, sitDBP<110mmHg
   * Blood pressure medication free patients: 140mmHg ≤ sitSBP<180mmHg, sitDBP<110mmHg
4. Visit2: 140mmHg ≤ sitSBP<180mmHg, sitDBP<110mmHg or if patients are in high risk group: 130mmHg ≤ sitSBP <180mmHg, sit DBP < 110mmHg

Exclusion Criteria:

* Difference in mean value of blood pressure measured in both arms of more than 20mmHg in sitSBP or more than 10mmHg in sitDBP
* Orthostatic hypotension with symptoms within 3months of visit 1
* Secondary hypertensive patient or suspected to be
* Uncontrolled diabetes mellitus(HbA1c > 9%) or type I diabetes mellitus
* Active gout or hyperuricemia (uric acid ≥ 9mg/dL)
* Severe heart disease or severe neurovascular disease
* Severe or malignant retinopathy
* Clinically significant hematological finding
* Severe renal diseases (eGFR<30mL/min/1.73m2)
* Severe hepatopathy or active hepatopathy (AST or ALT normal range ≥ 3 times)
* Hypokalemia or Hyperkalemia(K<3.5mmol/L or K ≥ 5.5mmol/L)
* Hyponatremia or Hypernatremia(Na<135mmol/L or Na ≥ 155mmol/L)
* Hypercalcemia
* History of malignancy tumor
* History of autoimmune disease
* History of alcohol or drug abuse
* Positive to pregnancy test, nursing mother, intention on pregnancy
* Considered by investigator as not appropriate to participate in the clinical study with othe reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean sitting systolic blood pressure(mmHg) | Week 8

SECONDARY OUTCOMES:
Change from baseline in mean sitting systolic blood pressure(mmHg) | Week 4
Change from baseline in mean sitting diastolic blood pressure(mmHg) | Week 4,8
Change from baseline in mean pulse blood pressure(mmHg) | Week 4,8
Responder rate | Week 4, 8
target blood pressure reach rate | Week 4, 8

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea